CLINICAL TRIAL: NCT00479531
Title: Sequential Compression Devices for Treatment of Restless Legs Syndrome - a Prospective, Randomized, Sham-Controlled Study
Brief Title: Sequential Compression Devices for Treatment of Restless Legs Syndrome
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Walter Reed Army Medical Center (U.S. Federal Agency)
Collaborators: AirCast LLC (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 05-17018
Record Dates: First submitted 2007-05-25; First posted 2007-05-28 (Estimated); Last update posted 2007-11-30 (Estimated); Status verified 2007-10

CONDITIONS: Restless Legs Syndrome
Keywords: Restless Legs Syndrome; Sequential Compression Device; Sleep Quality; Quality of Life
MeSH Terms: conditions — Restless Legs Syndrome; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: AirCast Sequential Compression Device

SUMMARY:
The purpose of this study is to determine if sequential compression devices (SCD) when worn for an hour per day by patients suffering from Restless Legs Syndrome (RLS) are helpful for the improvement of the RLS symptoms and sleep.

DETAILED DESCRIPTION:
Restless legs syndrome (RLS) is a highly vexing problem manifested by sensory and motor symptoms that disrupt sleep onset or sleep maintenance. RLS is the second most common sleep disorder and occurs with an estimated prevalence of 10% in the general population. The sleep disruption results in daytime symptoms such as excessive daytime sleepiness (EDS) and mood changes. There are no consistently reliable treatment alternatives. There is an urgent need for new, innovative treatment strategies because available pharmacological treatments often stop working over time or are associated with unacceptable side effects. An effective nonpharmacological treatment would be a highly attractive alternative.

Anecdotally, patients have reported that use of sequential compression devices (SCD) prescribed for prophylaxis of deep vein thrombosis can have a positive effect on RLS symptoms. Because this nonpharmacological alternative is available, safe, and affordable, further investigation is warranted.

Simply stated, the null hypothesis is that SCD therapy does not have an impact on RLS symptoms.

Patients will be randomized to wearing SCDs or sham SCDs for an hour each day prior to the usual onset of the RLS symptoms. At baseline and at monthly follow-ups for 3 to 4 months, participants will complete questionnaires to assess the severity of the RLS symptoms, their daytime sleepiness, and the impact of the RLS on quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 17 years with a reliable diagnosis of RLS in accordance with the International Classification of Sleep Disorders, Revised Diagnostic and Coding Manual of the American Academy of Sleep Medicine.

Exclusion Criteria:

* Age less than 18 years
* Unstable medical conditions that may interfere with the requirements of the study (for example uncontrolled diabetes mellitus, symptomatic asthma, congestive heart failure with symptoms of pulmonary edema), and mental or physical limitations (including dementia) that would preclude data collection on questionnaires or wearing the SCD.
* Other medical conditions that would serve as exclusion criteria are those where increased venous or lymphatic return is undesirable. These specific conditions are known or suspected acute deep vein thrombosis, thrombophlebitis, severe congestive heart failure, pulmonary edema, severe arteriosclerosis, active infection such as gangrene, recent vein ligation or skin graft, or extreme deformity of the legs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2005-09; Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Severity of RLS Symptom Score; Epworth Sleepiness Scale; Quality of Life Scores (RLS-QLI) | 3 to 4 months

SECONDARY OUTCOMES:
Compliance with SCD therapy by patient diary; Patient subjective experience by personal comments. | 3 to 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Lettieri, MD, Principal Investigator — Pulmonary & Critical Care Medicine Service, Walter Reed Army Medical Center, Washington DC
Locations (1):
- Christopher Lettieri MD, Sleep Disorders Center, Walter Reed Army Medical Center, District of Columbia, United States

REFERENCES:
- [Derived] Lettieri CJ, Eliasson AH. Pneumatic compression devices are an effective therapy for restless legs syndrome: a prospective, randomized, double-blinded, sham-controlled trial. Chest. 2009 Jan;135(1):74-80. doi: 10.1378/chest.08-1665. Epub 2008 Nov 18. PMID 19017878